CLINICAL TRIAL: NCT03981146
Title: A Phase II Trial Assessing Nivolumab in Class II Expressing Microsatellite Stable Colorectal Cancer
Acronym: ANICCA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-215; 2018-000318-39 (EudraCT Number); 40245896 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2019-05-09; First posted 2019-06-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: Class II Microsatellite Status
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Patients will receive 480mg of Nivolumab on a four weekly cycle for a maximum of two years.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — 60 Minute IV Infusion
  Other Names: Opdivo

SUMMARY:
An open-label, single-arm, phase II, multicentre clinical trial to determine the rate of durable clinical benefit of nivolumab in patients with class II expressing microsatellite stable colorectal cancer.

DETAILED DESCRIPTION:
Immuno-oncology is transforming the care of certain patients with cancer. Not all patients respond to these therapies however, and in some common cancers checkpoint blockade has failed to make any real impact. In 2014 there were over 41,000 new cases of colorectal cancer (CRC) in the UK and nearly 16,000 deaths from the disease, making it the second commonest cause of cancer death (Cancer Research UK Cancer Statistics Key Facts). 15% of patients with CRC develop it as a result of deficient mismatch repair (microsatellite instability - MSI): this cohort of patients respond well to PD-1/PD-L1 blockade as these tumours harbour a very high number of mutations thus increasing the likelihood of the presence of immunogenic neo-epitopes which elicit an immune response1. The majority of CRC patients, particularly those with metastatic disease (around 95%), do not display this hyper-mutator phenotype (microsatellite stable (MSS) CRC) and in these patients the results of PD-1/PD-L1 blockade have been disappointing.

In summary, MSS CRC patients with a class II expression appear to represent immunologically a group of MSI-like MSS patients that may respond to usefully to the immunotherapy agent nivolumab as a single agent and thus a trial of nivolumab in patients with class II expression of their cancer cells appears to be highly justified.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic MSS CRC with class II expression (greater than 1% cancer cell positivity for class II expression on immunohistochemistry).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (APPENDIX 1)
* Age ≥ 18 years
* Patients must have completed all standard of care therapy that the treating oncologist deems appropriate. Trial treatment as first line therapy is permitted if the patient has declined standard of care therapy.
* CT scan of chest, abdomen, pelvis within 28 days of registration demonstrating unidimensionally measurable disease as per RECIST version 1.1 (APPENDIX 3).
* Demonstrate adequate haematological function:

  * Platelet count ≥100 x 109 /L
  * Neutrophils ≥1.5 x 109/L
  * Haemoglobin ≥ 90 g/L
* Demonstrate adequate hepatic function:

  * Serum bilirubin ≤1.5 x upper limit of normal (ULN)
  * Serum AST or ALT ≤2.5 x ULN or <5 x ULN in the presence of liver metastases
* Demonstrate adequate renal function

  o Creatinine clearance <1.5 times ULN and >30ml/min (as per institutional standard).
* Provision of signed and dated, written informed consent prior to any trial specific procedures, sampling and analyses.
* Negative pregnancy test (female patients of reproductive potential). (Serum Test must be negative)
* Patients must agree to the use of contraception as detailed in section 7.8

Exclusion Criteria:

* Previous treatment with PD1/PDL1 inhibitors.

  * Untreated symptomatic brain or leptomeningeal metastatic disease.
  * Medical or psychiatric conditions compromising informed consent.
  * Any medical condition which, in the opinion of the Investigator, would compromise the ability of the patient to participate in the trial or which would jeopardise compliance with the protocol.
  * Administration of chemotherapy, radioactive or biological cancer therapy within 4 weeks prior to the first dose of trial therapy Patient has not recovered to CTCAE grade 1 or better from the Adverse Event (AE) due to cancer therapeutics administered more than 4 weeks earlier.
  * Active autoimmune disease that has required systemic treatment in past 2 years (i.e.

with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patient has risk factors for bowel obstruction or bowel perforation (examples include but not limited to a history of acute diverticulitis, intra-abdominal abscess and abdominal carcinomatosis).
* Patient has a known history of other malignancy, unless the patient has undergone potentially curative therapy with no evidence of that disease for 3 years.
* Has a history of non-infectious pneumonitis requiring steroids or has active pneumonitis.
* Female patients that are either pregnant or breast feeding.
* Male and female patients (of childbearing age) not willing to use adequate contraception.
* Patient previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Patient is positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA (qualitative) is detected); patients with negative Hepatitis C antibody testing may not need RNA testing.
* Known history of tuberculosis.
* Patient has an active infection requiring therapy.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Durable Clinical Benefit | Beginning of trial treatment to free of disease progression (104 weeks maximum)
  patient will be defined as experiencing DCB if they remain free of disease progression at their third trial specific CT scan since treatment start date (i.e. at approximately 27 weeks) or at any CT scan after 27 weeks that shows the patient remains free of disease progression

SECONDARY OUTCOMES:
Objective response | trial treatment until disease progression (104 weeks maximum)
  Objective response is the occurrence of CR or PR as the best overall response
Best Percentage Change in Sum of Target Lesions | Trial Treatment to disease progression (104 weeks maximum)
  At each evaluation, the longest diameters of all selected target lesions will be measured and summed and the percentage change from the baseline measurement will be calculated. The best percentage change is the one that reflects either the greatest decrease or the least increase over the whole period of assessment.
Time to Maximal Response | Occurrence of CR or PR during the trial (104 weeks maximum)
  This is defined as the time from commencement of trial treatment to the date of CT scan that first records the best objective response as per RECIST version 1.1.
Progression Free Survival Time | time from commencement of trial treatment to the date of CT scan when progressive disease first recorded (104 weeks maximum)
  This is defined as the time from commencement of trial treatment to the date of CT scan when progressive disease first recorded or date of death without previously recorded progression.first records the best objective response as per RECIST version 1.1.
Overall Survival Time | Trial Treatment to date of death.
  This is defined as the time from commencement of trial treatment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Middleton, MB,BS,FRCP, Principal Investigator — University of Birmingham
Locations (14):
- United Kingdom (14):
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - St James Leeds, Leeds
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - The Royal Free Hospital, London
  - Guys Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College Hospital, London
  - The Christie Hospital, The Christie NHS Foundation Trust, Manchester
  - Freemans Hospital, Newcastle upon Tyne
  - Weston Park, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial Website — https://www.birmingham.ac.uk/research/crctu/trials/Anicca-classII/ANICCA-Class-II.aspx